CLINICAL TRIAL: NCT01860040
Title: Neoadjuvant Chemotherapy for Non-metastatic Non-small Cell Lung Cancer
Brief Title: Neoadjuvant Chemo for Non-metastatic Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual, no data to analyze
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-04
Record Dates: First submitted 2013-05-17; First posted 2013-05-22 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Non-squamous Cell Non-Metastatic Non-Small Cell Lung Cancer; Squamous Cell Non-Metastatic Non-Small Cell Lung Cancer
MeSH Terms: interventions — Cisplatin; Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cisplatin and pemetrexed (Experimental): Cisplatin on day 1 and pemetrexed on day 1, 1 cycle = 21 days, deliver 4 neoadjuvant cycles
  Interventions: Drug: Cisplatin; Drug: Pemetrexed
- Cisplatin and gemcitabine (Experimental): Cisplatin on day 1 and gemcitabine on days 1 and 8, 1 cycle = 21 days, deliver 4 neoadjuvant cycles
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Cisplatin — Alkylating antineoplastic agent (Chemotherapy)
  Other Names: Platinol®
Drug: Pemetrexed — Antimetabolite antineoplastic agent (Chemotherapy)
  Other Names: Alimta®
  Arms: Cisplatin and pemetrexed
Drug: Gemcitabine — Antimetabolite antineoplastic agent (Chemotherapy)
  Other Names: Gemzar®
  Arms: Cisplatin and gemcitabine

SUMMARY:
To determine the rate of pathologic complete responses (pCR) at the time of definitive surgical resection of non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
Participants in this study will have a lung mass and are undergoing a procedure to determine if they have non-small cell lung cancer that could be removed surgically. If confirmed to have non-small cell lung cancer that can be surgically removed, he or she may be able to continue as a possible participant in this study.

The purpose of this study is to determine whether neoadjuvant chemotherapy (chemotherapy that is given before surgery) will improve the amount of time a participant is free from disease in people with non-metastatic (has not spread from the original site) non-small cell lung cancer. The chemotherapy medications that will be used in this study are cisplatin and pemetrexed or cisplatin and gemcitabine and have been shown to be effective in patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age with either a mass suspicious for or histologically confirmed AJCC stage IB-IIIA NSCLC. For those without histologic confirmation of NSCLC, a biopsy will be done and only those patients with histologically confirmed NSCLC meeting all other eligibility criteria may proceed on protocol.
2. Mass must be determined to be surgically resectable
3. Eastern Cooperative Oncology Group (ECOG) performance status score < 1 and a life expectancy >3 months.
4. Participants must have at least one evaluable lesion as defined by RECIST 1.1
5. Absolute neutrophil count > 1500 mm3, platelet count ≥ 100×109 L, hemoglobin ≥ 8.5 g/dL
6. Serum creatinine ≤1.3 mg/dL (candidate for cisplatin chemotherapy), total bilirubin ≤ 2 mg/dL, AST/ALT ≤ 5 times the upper limit of normal range
7. No prior chemotherapy or radiotherapy for NSCLC
8. At least 5 years from diagnosis of another cancer except treated in-situ disease or surgically resected non-melanoma skin cancer with clear margins.
9. Willingness to provide permission to biopsy NSCLC for collection of frozen pretreatment sample.
10. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable contraceptive method (abstinence, oral contraceptive or double barrier method) for the duration of the study and for 30 days following the last dose of study drug, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial

Exclusion Criteria:

1. Active clinically serious infection > CTCAE (version 4.03) Grade 2.
2. Serious non-healing wound, ulcer, or bone fracture.
3. Major contraindication to surgical resection of NSCLC
4. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements.
5. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements.
6. Patients receiving any other investigational agents.
7. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen Weiss, MD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: did not meet recruitment goal
Groups:
- Cisplatin and Pemetrexed: Cisplatin on day 1 and pemetrexed on day 1, 1 cycle = 21 days, deliver 4 neoadjuvant cycles
  Cisplatin
  Pemetrexed
- Cisplatin and Gemcitabine: Cisplatin on day 1 and gemcitabine on days 1 and 8, 1 cycle = 21 days, deliver 4 neoadjuvant cycles
  Cisplatin
  Gemcitabine
Period: Overall Study
Arm/Group | Cisplatin and Pemetrexed | Cisplatin and Gemcitabine
Started | 1 (did not meet recruitment goal) | 0 (did not meet recruitment goal)
Completed | 0 (did not meet recruitment goal) | 0 (did not meet recruitment goal)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisplatin and Pemetrexed | Cisplatin and Gemcitabine | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Pathologic Complete Responses (pCR) at the Time of Definitive Surgical Resection of Non-small Cell Lung Cancer
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by Magnetic Resonance Imagery (MRI): Complete Response (CR), Disappearance of all target lesions
Time Frame: One year
Population: There are no data recordings for this study. The study was terminated and the investigator is no longer related to the site. There is no additional information to provide.
Arm/Group | Cisplatin and Pemetrexed
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cisplatin and Pemetrexed | Cisplatin and Gemcitabine
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin and Pemetrexed (N=1) | Cisplatin and Gemcitabine (N=0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin and Pemetrexed (N=1) | Cisplatin and Gemcitabine (N=0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes